CLINICAL TRIAL: NCT01872078
Title: A Randomised, Double-blind, Placebo-controlled Phase IIa Study to Assess the Pharmacodynamics, Safety, and Pharmacokinetics of AZD4901 When Given in Multiple Doses to Females With Polycystic Ovary Syndrome
Brief Title: A Study of AZD4901 in Females With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5320C00001
Record Dates: First submitted 2013-05-23; First posted 2013-06-07 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Polycystic Ovary Syndrome (PCOS), Female Endocrine Disorder
Keywords: Pharmacokinetics, Pharmacodynamics, endocrinopathies, PCOS, female, hormone, LH
MeSH Terms: conditions — Polycystic Ovary Syndrome; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD4901 20 mg once a day (Experimental): AZD4901 20 mg once a day
  Interventions: Drug: AZD4901 (oral)
- AZD4901 20mg twice a day (Experimental): AZD4901 20mg twice a day
  Interventions: Drug: AZD4901 (oral)
- AZD4901 40 mg twice a day (Experimental): AZD4901 40 mg twice a day
  Interventions: Drug: AZD4901 (oral)
- Placebo to match AZD4901 (Experimental)
  Interventions: Drug: Placebo to match AZD4901

INTERVENTIONS:
Drug: AZD4901 (oral) — Patients randomized to 1 of 4 treatment groups: AZD4901 20 mg once a day, AZD4901 20 mg twice a day, AZD4901 40 mg twice a day or placebo
  Arms: AZD4901 20 mg once a day; AZD4901 20mg twice a day; AZD4901 40 mg twice a day
Drug: Placebo to match AZD4901 — Patients randomized to 1 of 4 treatment groups: AZD4901 20 mg once a day, AZD4901 20 mg twice a day, AZD4901 40 mg twice a day or placebo
  Arms: Placebo to match AZD4901

SUMMARY:
To assess the effects of AZD4901 when given in multiple doses to females with Polycystic Ovary Syndrome

ELIGIBILITY:
Inclusion Criteria:

Female patients between the ages of 18 to 45 years (inclusive). Suitable veins for cannulation or repeated venipuncture. Body mass index (BMI) between 18 and 40 kg/m2 (inclusive). A diagnosis of polycystic ovary disease. Amenorrhea or oligomenorrhea (defined as ≤ 6 menses per year). Negative serum pregnancy test at screening. Negative urine pregnancy test before randomisation. Not be breast-feeding. Not have been pregnant within the 6 months prior to screening.

Exclusion Criteria:

Perimenopausal or reached natural menopause, defined as FSH > 10 IU/L. Menstruated within the month prior to the baseline visit. Hysterectomy or bilateral oophorectomy or both. Clinically relevant disease and abnormalities (past or present), and in particular causes of abnormal vaginal bleeding.

Withdrawals from oral contraceptives if their LH levels are below 3 IU/L when retested within 7 ± 1 days of the baseline visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyothis George, MD, Principal Investigator — University of Oxford
Locations (7):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Springfield, Missouri
- Research Site, Berlin, Germany
- United Kingdom (3):
  - Research Site, Belfast
  - Research Site, Edinburgh
  - Research Site, London

REFERENCES:
- [Derived] George JT, Kakkar R, Marshall J, Scott ML, Finkelman RD, Ho TW, Veldhuis J, Skorupskaite K, Anderson RA, McIntosh S, Webber L. Neurokinin B Receptor Antagonism in Women With Polycystic Ovary Syndrome: A Randomized, Placebo-Controlled Trial. J Clin Endocrinol Metab. 2016 Nov;101(11):4313-4321. doi: 10.1210/jc.2016-1202. Epub 2016 Jul 26. PMID 27459523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 patients were recruited to the study, of which 65 received doses of AZD4901 between 20 mg qd and 40 mg bid or placebo. Two patients were excluded due to poor venous access
Groups:
- Placebo: Two matching placebo tablets for both the morning and evening doses
- 20 mg AZD4901 Once Daily: One 20-mg AZD4901 tablet and 1 placebo tablet for the morning dose and 2 placebo tablets for the evening dose
- 20 mg AZD4901 Twice Daily: One 20-mg AZD4901 tablet and 1 placebo tablet for both the morning and evening doses
- 40 mg AZD4901 Twice Daily: Two 20-mg AZD4901 tablets for both the morning and evening doses
Period: Overall Study
Arm/Group | Placebo | 20 mg AZD4901 Once Daily | 20 mg AZD4901 Twice Daily | 40 mg AZD4901 Twice Daily
Started | 16 | 15 | 17 | 17
Completed | 16 | 15 | 14 | 15
Not Completed | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Dose administration non-compliance | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Patient met exclusion criterion 16. | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 20 mg AZD4901 Once Daily | 20 mg AZD4901 Twice Daily | 40 mg AZD4901 Twice Daily | Total
Number analyzed (Participants) | 16 | 15 | 17 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27 (3) | 29 (6) | 27 (6) | 28 (6) | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 17 | 17 | 65
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lutenising Hormone (LH) AUC(0-8) Ratio to Baseline at Day 7
Description: Change-from-baseline of luteinising hormone area under the concentration-time curve from time zero to 8 hours postdose [AUC(0-8)] at Day 7
Time Frame: Day 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- 20 mg AZD4901 qd: 20 mg AZD4901 once daily administered orally
- 20 mg AZD4901 Bid: 20 mg AZD4901 twice daily administered orally
- 40 mg AZD4901 Bid: 40 mg AZD4901 twice daily administered orally
Arm/Group | Placebo | 20 mg AZD4901 qd | 20 mg AZD4901 Bid | 40 mg AZD4901 Bid
Number analyzed (Participants) | 13 | 13 | 14 | 15
Ratio | 1.118 [0.8446 to 1.479] | 0.9729 [0.7351 to 1.288] | 0.8804 [0.6724 to 1.153] | 0.5364 [0.4134 to 0.6960]
Statistical Analysis 1: Comparison: Placebo vs 20 mg AZD4901 qd; The null hypothesis is that the ratio of Active to Control in LH AUC(0-8) ratio to baseline at day 7= 100%; Test type: Superiority or Other; Ratio (%) = 87.04, 95% CI 2-sided [58.52 to 129.47]
Statistical Analysis 2: Comparison: Placebo vs 20 mg AZD4901 Bid; The null hypothesis is that the ratio of Active to Control in LH AUC(0-8) ratio to baseline at day 7= 100%; Test type: Superiority or Other; Ratio (%) = 78.76, 95% CI 2-sided [53.41 to 116.16]
Statistical Analysis 3: Comparison: Placebo vs 40 mg AZD4901 Bid; The null hypothesis is that the ratio of Active to Control in LH AUC(0-8) ratio to baseline at day 7= 100%; Test type: Superiority or Other; Ratio (%) = 47.99, 95% CI 2-sided [32.73 to 70.36]

ADVERSE EVENTS:
Arm/Group | 20 mg AZD4901 Once Daily | 20 mg AZD4901 Twice Daily | 40 mg AZD4901 Twice Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 6/15 | 13/17 | 5/17 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg AZD4901 Once Daily (N=15) | 20 mg AZD4901 Twice Daily (N=17) | 40 mg AZD4901 Twice Daily (N=17) | Placebo (N=16)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 20 mg AZD4901 Once Daily (N=15) | 20 mg AZD4901 Twice Daily (N=17) | 40 mg AZD4901 Twice Daily (N=17) | Placebo (N=16)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0/0 | 1/1 | 0/0 | 0/0
Tooth fracture (Injury, poisoning and procedural complications) | 0/0 | 1/1 | 0/0 | 0/0
Headache (Nervous system disorders) | 2 | 3 | 4 | 5
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 2 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca will manage the publication of the results of the Clinical Trial in partnership with the authors. AstraZeneca recognises that Institutions/Investigators may wish to make publications regarding Clinical Trial results. The Institution/Investigator agrees to collaborate in good faith with AstraZeneca. Prior to any such publication, the Institution/Investigator shall provide AstraZeneca with preliminary data and drafts of proposed publications.